CLINICAL TRIAL: NCT06561204
Title: Impact of a Full-mouth Electronic Toothbrush on Indicators of Gingivitis and Patient Perceptions: A Randomized Clinical Trial
Brief Title: Full-mouth Electronic Toothbrush vs. Conventional Electronic Toothbrush
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: FENO.Co (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00022906
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Toothbrush; Gingivitis; Plaque
MeSH Terms: conditions — Gingivitis; Plaque, Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FMET + ADA dentifrice (Experimental): Baseline and 30-day outcome measures will be collected to evaluate the impact of FMET + ADA dentifrice on clinical indicators of gingivitis, plaque, and patient perceptions.
  Interventions: Device: FMET
- Conventional electronic toothbrush + ADA dentifrice (No Intervention): Baseline and 30-day outcome measures will be collected to evaluate the impact of conventional electronic toothbrush + ADA dentifrice on clinical indicators of gingivitis, plaque, and patient perceptions.
- FMET + Foam (Other): Baseline and 30-day outcome measures will be collected to evaluate the impact of FMET + foam on clinical indicators of gingivitis, plaque, and patient perceptions.
  Interventions: Device: FMET

INTERVENTIONS:
Device: FMET — A full-mouth electronic toothbrush
  Arms: FMET + ADA dentifrice; FMET + Foam

SUMMARY:
The goal of this randomized, masked-examiner clinical trial is to investigate a full-mouth electronic toothbrush (FMET). The three arms are: 1) FMET + American Dental Association (ADA) approved dentifrice, 2) conventional electronic toothbrush (ETB) + ADA dentifrice and 3) FMET + foam system.

DETAILED DESCRIPTION:
The primary purpose is to compare the FMET + ADA dentifrice to the conventional ETB + ADA dentifrice. The exploratory aim is to compare the FMET + foam system to both the FMET + ADA dentifrice and conventional ETB + ADA dentifrice. Baseline and 30-day outcome measures will be collected to evaluate the impact on clinical indicators of gingivitis, plaque, and patient perceptions.

ELIGIBILITY:
Inclusion Criteria:

* University of Minnesota School of Dentistry patient of record who is 18 years of age or older.
* Documented periodontal classification of mild to moderate gingivitis (>10% BOP) or documented gingivitis on an intact, reduce, or stable with a history of periodontitis in AxiUm electronic health record (EHR) >10% BOP.
* A minimum of 25% plaque measured O'Leary plaque score.
* A minimum of five natural teeth in each quadrant (excluding third molars, dental implants or teeth with more that ½ of natural surface restored).
* Be willing to abstain from all professional oral hygiene care (prophy/periodontal maintenance) during the study.
* Be willing to abstain from the use of any other dental cleaning aids (dental floss, water flossers, interdental brushes, dental or tooth picks, mouthwash, etc.) during the study.
* Access to personal email account and a device connected to the internet to complete questionnaires and communicate with study team.

Exclusion Criteria:

* Presence of aggressive, necrotizing, uncommon periodontal disease, or any uncontrolled periodontal condition.
* Presence of any physical limitation or restriction that might preclude normal oral hygiene procedures (i.e. need another individual to perform oral self-care).
* Fixed prosthesis (i.e. implant retained denture), orthodontic appliance or under orthodontic treatment.
* Any medication that may impact periodontal conditions (i.e., phenytoin, calcium antagonists, cyclosporin, warfarin, antimicrobials, or steroids).
* Have any uncontrolled medical condition or immunocompromised that may impact the study (i.e. uncontrolled diabetes HbA1c > 7, HIV).
* Pregnant, planning to become pregnant, or unsure of pregnancy status (self-reported)
* ≥2 weeks of antibiotic use in the past three months. Or antibiotic use in the last six weeks.
* Cigarette use within the last year
* Unable to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Löe & Silness gingival index (GI) | Baseline and 30-days
  Scale 0-3
Turesky modification of the Quigley-Hein index | Baseline and 30-days
  Scale 0-5

CONTACTS AND LOCATIONS:
Overall Officials: Michelle C Arnett, MS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota School of Dentistry, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers.